CLINICAL TRIAL: NCT04625114
Title: The Potential of Oral Camostat in Early COVID-19 Disease in an Ambulatory Setting to Reduce Viral Load and Disease Burden
Brief Title: The Potential of Camostat in COVID-19
Acronym: COV-AAT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analyses did not show evidence that camostat mesylate under the present conditions (300 mg three times daily for five or 10 consecutive days, fasted state) was effective as an antiviral drug against early phase SARS-CoV-2 disease.
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BC-7707
Record Dates: First submitted 2020-11-05; First posted 2020-11-12 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Covid19
Keywords: antiviral
MeSH Terms: conditions — COVID-19 | interventions — camostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: double blinded placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Camostat (Experimental): camostat 100mg 3 tablets 3x/day D1->D5 (+ possible extension D6->D10)
  Interventions: Drug: Camostat
- Placebo (Placebo Comparator): Placebo 3 tablets 3x/day D1->D5 (+ possible extension D6->D10)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Camostat — Standard of care (SOC) + Camostat mesilate (Foipan) 100mg 3 tablets 3 times a day for 5 consecutive days (D1->D5);
  Arms: Camostat
Drug: Placebo — SOC + placebo 500 mg 3 tablets 3 times a day for five consecutive days (D1->D5).
  Arms: Placebo
Drug: Camostat — Standard of care (SOC) + Camostat mesilate (Foipan) 100mg 3 tablets 3 times a day for 5 consecutive days (D6->D10);
  Arms: Camostat
Drug: Placebo — SOC + placebo 500 mg 3 tablets 3 times a day for five consecutive days (D6->D10).
  Arms: Placebo

SUMMARY:
The investigators are conducting a pilot trial where they will study safety, efficacy and compliance in a cohort of ambulatory patients in the Ghent region with confirmed COVID-19 infection, in both an early stage of disease, defined as less than 5 days of symptoms and who at presentation do not meet any criteria for hospitalisation as well as asymptomatic individuals with a PCR CT value below 30.

The primary endpoint is to assess the efficacy of the drug in terms of change from day 0 to day 5 in respiratory (oropharyngeal swab RT-PCR) log10 viral load.

The aim of the study is to assess whether Camostat, a serine protease inhibitor available in an oral formulation has the potential to be studied as an antiviral drug in a large scale ambulatory setting to prevent transmission by decreasing viral load, to prevent symptoms after exposure (PEP) in asymptomatic individuals or to prevent disease progression in the occurrence of early symptomatology.

DETAILED DESCRIPTION:
Core study After eligibility assessment participants will be randomized and will receive the study drugs. We will define D1 as the first dose of the medication which can be the morning, midday or evening dose. They will be treated for 5 consecutive days.

In patients with a positive PCR at D5 (CT value with threshold below 30) and/or presence of clinical symptoms after exclusion of hospitalization criteria (flowchart emergency department appendix 4), the treatment will be extended up to D10 at the same dosage in both treatment arms for 5 consecutive days: D6 and D10).

Follow-up will be as follows:

* D1->D14 (D28): The study participants will be asked to fill in daily questionnaires assessing symptoms (cfr daily self-score). They will receive a kit enabling to monitor heart rate (HR), respiratory rate (RR), temperature and oxygen saturation 3 times per day (every 4-8 hours, preferentially at the timing of medication intake at D1 to D5 or D10).
* Compliance and tolerance will be assessed during the treatment period, D0->D5 (or D0->D10 if the treatment is prolonged).
* During the study D1-D28: If indicated in the opinion of the investigator, a physical exam and biochemistry will be performed through a consultation at the clinic. This can be requested at any time during the study based on clinical symptoms or signs.
* Consultation at D0, D5, (D10) and D28 at our COVID consultation facility. This will be done by a study nurse and/or a study physician.

ELIGIBILITY:
Inclusion Criteria

* Aged ≥18
* Willing to participate and fill out a daily symptom diary
* Willing to take the parameters such as blood oxygenation and temperature
* Willing to attend follow-up visits both by phone as at the clinic
* Capable of understanding the commitment in the trial
* Signed informed consent
* Signs and symptoms suggestive of COVID disease in absence of hospitalization criteria as defined by the flowchart used at the emergency department of our institution (appendix 4), present for maximum 5 days and confirmed by PCR.
* OR documented COVID-19 infection by PCR with CT value below the threshold of 30 in asymptomatic individuals.
* For women of childbearing potential*: they should be willing to use highly effective method of contraception during treatment and until the end of study defined as having a failure rate of less than 1% per year when used consistently and correctly.

Such methods include:

* combined (estrogen and progestogen containing) hormonal contraception
* associated with inhibition of ovulation: oral, intravaginal or transdermal
* progestogen-only hormonal contraception associated with inhibition of ovulation: oral, injectable or implantable
* intrauterine device (IUD) and intrauterine hormone-releasing system ( IUS)
* bilateral tubal occlusion
* vasectomised partner
* sexual abstinence

  * For men of reproductive potential**: condom should be used as contraception during treatment and until the end of study when having a partner of childbearing potential

    * a woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.

      * a man is considered fertile after puberty unless permanently sterile by bilateral orchidectomy.

Exclusion Criteria

* Inability to make a decision to participate
* Pregnant or breast feeding
* Inability to take oral medication
* Inability to provide informed written consent
* Known hypersensitivity towards Camostat or other Serine protease inhibitors
* Any condition that, in the Investigator's opinion, prevents adequate compliance with study therapy.
* Any COVID infection at risk for hospitalisation as described in the emergency department flowchart (cfr appendix 4)
* With regard to exclusion of women of child-bearing potential, women who tell us they know they are pregnant are excluded. All women of child-bearing potential who test positive for pregnancy by urine test at first visit are excluded.
* Severe chronic pancreatitis requiring suction of gastric juice, fasting or abstention from drinking
* Postoperative reflux oesophagitis due to reflux or gastric juice
* Postoperative reflux oesophagitis (if improvement of symptoms is not observed).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Callens, Principal Investigator — UZ Gent
Locations (1):
- Ghent University Hospital, Algemene Inwendige Ziekten, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tobback E, Degroote S, Buysse S, Delesie L, Van Dooren L, Vanherrewege S, Barbezange C, Hutse V, Romano M, Thomas I, Padalko E, Callens S, De Scheerder MA. Efficacy and safety of camostat mesylate in early COVID-19 disease in an ambulatory setting: a randomized placebo-controlled phase II trial. Int J Infect Dis. 2022 Sep;122:628-635. doi: 10.1016/j.ijid.2022.06.054. Epub 2022 Jul 5. PMID 35803469

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Camostat | Placebo
Started | 66 | 30
Initial Treatment Period (D1-D5) | 52 | 25
Extension Needed (D6-D10) | 9 | 4
Completed | 61 | 29
Not Completed | 5 | 1
Not completed — Adverse Event | 3 | 1
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: Between Nov2020 and Jun2021, a total of 108 participants were enrolled in the study. 12 subjects did not meet the in- and exclusion criteria and were excluded from randomization. A total of 96 participants received either camostat (N=66) or placebo (N=30). Treatment was interrupted in 4 subjects that had to be hospitalized due to clinical deterioration. Two other subjects chose to withdraw from the study. Analyses were performed on the data of 90 participants who completed treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Camostat | Placebo | Total
Number analyzed (Participants) | 61 | 29 | 90
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 38 [25 to 53] | 37 [22 to 51] | 38 [25 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 16 | 49
  Male | 28 | 13 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 59 | 29 | 88
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Belgium | 61 | 29 | 90

OUTCOME MEASURES:

1. Primary Outcome: Efficacy in Terms of Viral Load or Surrogate After 5 Days of Treatment
Description: The primary endpoint is to assess the efficacy of the drug in terms of change from day 0 to day 5 in respiratory (oropharyngeal swab RT-PCR) surrogate market CT value. Higher values equate to better outcomes.
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: number of cycles
Arm/Group | Camostat | Placebo
Number analyzed (Participants) | 61 | 29
number of cycles | 2.34 (10.27) | 2.08 (11.14)
Statistical Analysis 1: Comparison: Camostat vs Placebo; Test type: Superiority; p = 0.511, Mixed Models Analysis; Mean Difference (Final Values) = 1.183

2. Secondary Outcome: Number of Patients With Clinical Improvement (in at Least 1 Point on the 5-point Likert Scale) of 5 Most Self-reported Symptoms
Description: Symptoms were daily measured by means of a self-report questionnaire. The top 5 self-reported symptoms during the whole study period were determined. Time to clinical improvement of these 5 most self-reported symptoms were compared between the camostat and placebo group. Additionally, potential risk factors are studied in order to influence clinical improvement.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Camostat | Placebo
Number analyzed (Participants) | 61 | 29
Participants | 22 | 13
Statistical Analysis 1: Comparison: Camostat; Test type: Superiority; p = 0.921, Regression, Cox; Cox Proportional Hazard = 0.965, 95% CI 2-sided [0.480 to 1.942]

3. Secondary Outcome: Neutralizing Antibodies (NAbs) at Visit 28
Description: The 50% neutralizing antibody titer (NT50) was compared between the camostat and placebo group
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Camostat | Placebo
Number analyzed (Participants) | 61 | 29
Participants
  NT50 higher than the detection limit (≥40) | 38 | 22
  NT50 below the detection limit (<40) | 23 | 7

ADVERSE EVENTS:
Time Frame: adverse events were recorded from the time the subject has taken at least one dose of study treatment (day 1) through the last visit of this subject (day 28 visit).
Description: Patients were selected either based on the presence of symptoms suggestive of COVID-19 disease based on clinical symptoms and signs or any asymptomatic individual that presented with positive screening test. Patients that needed to be hospitalized or had a high risk of hospitalization were not included.
Arm/Group | Camostat | Placebo
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/29
Serious Adverse Events (participants affected / at risk) | 3/61 | 1/29
Other Adverse Events (participants affected / at risk) | 59/61 | 23/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Camostat (N=61) | Placebo (N=29)
COVID-19 pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) — 4 participants were hospitalized, because of severe COVID-19 pneumonia (1), mild to moderate COVID-19 pneumonia (1), deterioration of COVID-19 disease (1), COVID-19 pneumonia and exhaustion (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Camostat (N=61) | Placebo (N=29)
fatigue (General disorders) | 19 | 4
change in appetite (Metabolism and nutrition disorders) | 9 | 2
diarrhea (Gastrointestinal disorders) | 7 | 4
nausea (Gastrointestinal disorders) | 9 | 2
headache (Nervous system disorders) | 5 | 2
flatulence (Gastrointestinal disorders) | 4 | 0
dizziness (Ear and labyrinth disorders) | 3 | 0
neutropenia (Investigations) | 9 | 2
leucopenia (Investigations) | 7 | 2
CRP increase (Investigations) | 4 | 2
lymphopenia (Investigations) | 4 | 2
ALT increase (Investigations) | 3 | 2
ferritin increase (Investigations) | 3 | 2
fibrin D dimer increase (Investigations) | 3 | 2
eosinopenia (Investigations) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-04): https://cdn.clinicaltrials.gov/large-docs/14/NCT04625114/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-04): https://cdn.clinicaltrials.gov/large-docs/14/NCT04625114/ICF_001.pdf